CLINICAL TRIAL: NCT01234857
Title: A Two-Part Adaptive, Randomized Trial of Ridaforolimus in Combination With Dalotuzumab Compared to Exemestane or Compared to Ridaforolimus or Dalotuzumab Monotherapy in Estrogen Receptor Positive Breast Cancer Patients
Brief Title: A Study of Ridaforolimus (MK-8669) in Combination With Dalotuzumab (MK-0646) Compared to Standard of Care Treatment in Estrogen Receptor Positive Breast Cancer Patients (MK-8669-041 AM3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-041
Record Dates: First submitted 2010-09-22; First posted 2010-11-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: mTOR; breast cancer; estrogen receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — ridaforolimus; dalotuzumab; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A: ridaforolimus + dalotuzumab (Experimental): Approximately 15 patients will be enrolled to the ridaforolimus-dalotuzumab combination treatment arm. Subsequent Patients are randomly assigned in a 1:1 ratio to treatment with the ridaforolimus (20 mg daily five days a week)/dalotuzumab (intravenous infusion 10 mg/kg once weekly) combination therapy or cross-over to exemestane single-therapy treatment.
  Interventions: Drug: ridaforolimus + dalotuzumab
- Part A: exemestane (Active Comparator): Exemestane 25 mg daily; single-agent therapy.
  Interventions: Drug: exemestane
- Part B: ridaforolimus + dalotuzumab (Experimental): Patients are randomly assigned in a 1:1 ratio to treatment with the ridaforolimus (20 mg daily five days a week)/dalotuzumab (intravenous infusion 10 mg/kg once weekly) combination therapy or cross-over to one of two single-therapy treatments (ridaforolimus alone or dalotuzumab alone). With the implementation of Amendment 3, this study arm will not be opened.
  Interventions: Drug: ridaforolimus + dalotuzumab
- Part B: ridaforolimus (Experimental): Ridaforolimus; 40 mg daily five days a week, single-agent therapy. With the implementation of Amendment 3, this study arm will not be opened.
  Interventions: Drug: ridaforolimus
- Part B: dalotuzumab (Experimental): Dalotuzumab intravenous infusion 10 mg/kg weekly; single-agent therapy. With the implementation of Amendment 3, this study arm will not be opened.
  Interventions: Drug: dalotuzumab

INTERVENTIONS:
Drug: ridaforolimus + dalotuzumab — Ridaforolimus 20 mg once daily (QD) five days a week, with the possibility of escalation to 30 mg once daily (QD) after the first cycle and dalotuzumab intravenous infusion 10 mg/kg once weekly (QW). Treatment will continue until disease progression.
  Other Names: MK-8669, MK-0646
  Arms: Part A: ridaforolimus + dalotuzumab; Part B: ridaforolimus + dalotuzumab
Drug: exemestane — Exemestane 25 mg daily (QD). Treatment will continue until disease progression. Patients may cross-over to the combination therapy after disease progression at the discretion of the investigator with Sponsor approval.
  Arms: Part A: exemestane
Drug: ridaforolimus — Ridaforolimus 40 mg QD five days a week. Treatment will continue until disease progression. Patients may cross-over to the combination therapy after disease progression at the discretion of the investigator with Sponsor approval. Note: the Sponsor-recommended dose of ridaforolimus when administered as a single agent is 40 mg/day, but when given in combination with dalotuzumab, it is given at 30 mg/day.
  Other Names: MK-8669
  Arms: Part B: ridaforolimus
Drug: dalotuzumab — Dalotuzumab intravenous infusion 10 mg/kg QW. Treatment will continue until disease progression. Patients may cross-over to the combination therapy after disease progression at the discretion of the investigator with Sponsor approval.
  Other Names: MK-0646
  Arms: Part B: dalotuzumab

SUMMARY:
This is a two-part study that will determine, if: 1) the combination of ridaforolimus and dalotuzumab will improve progression-free survival compared to exemestane; and 2) the combination of ridaforolimus and dalotuzumab will improve progression-free survival compared to both ridaforolimus and dalotuzumab as single agents, in participants with breast cancer.

ELIGIBILITY:
Inclusion Criteria The prospective participant must meet, at least, all of the criteria below to be eligible for study participation.

The participant:

* Has a confirmed diagnosis of breast cancer that is metastatic or locally advanced and is estrogen receptor positive and human epidermal growth factor receptor 2 (HER-2) negative ;
* Is post-menopausal;
* Is at least 18 years of age;
* Has a life expectancy of at least 3 months;
* Has had a recurrence or progression of cancer after prior treatment and patient has received at least one line of endocrine therapy for metastatic disease, OR the patient's cancer has recurred within 6 months after the last dose of anastrozole or letrozole;
* Has an available archival tumor specimen;
* Has voluntarily agreed to participate by signing informed consent.

Exclusion Criteria If the prospective participant meets any of the criteria below (among others determined by the study staff) they will NOT be eligible for study participation.

The participant:

* Is receiving any other systemic tumor therapy;
* Has previously received rapamycin or rapamycin analogs;
* Has received prior treatment with insulin-like growth factor 1 receptor (IGF-1R) inhibitors, phosphoinositide 3-kinase (PI3K) inhibitors, or other experimental agents that target the PI3K, protein kinase B (AKT), or mammalian target of rapamycin (mTOR) pathways;
* Has known allergy to macrolide antibiotics;
* Has an active infection that requires antibiotics;
* Has significant or uncontrolled cardiovascular disease;
* Has poorly controlled Type 1 or 2 diabetes mellitus;
* Is known to be human immunodeficiency virus (HIV) positive;
* Has a known history of active Hepatitis B or C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-09-17 (Actual); Primary Completion 2013-10-15 (Actual); Study Completion 2013-10-15 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Assessed every 8 weeks until documentation of disease progression or death.
  Progression free survival is defined as the time from randomization to progressive disease or death, which ever occurs earlier.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Assessed every 8 weeks until documentation of disease progression or death.
  Objective response rate (ORR) will be estimated by the proportion of patients who achieve partial response (PR) or complete response (CR) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Overall survival (OS) | Every 3 months after participants go off active treatment
  Overall survival is defined as the time from randomization to death due to any cause.

REFERENCES:
- [Result] Baselga J, Morales SM, Awada A, Blum JL, Tan AR, Ewertz M, Cortes J, Moy B, Ruddy KJ, Haddad T, Ciruelos EM, Vuylsteke P, Ebbinghaus S, Im E, Eaton L, Pathiraja K, Gause C, Mauro D, Jones MB, Rugo HS. A phase II study of combined ridaforolimus and dalotuzumab compared with exemestane in patients with estrogen receptor-positive breast cancer. Breast Cancer Res Treat. 2017 Jun;163(3):535-544. doi: 10.1007/s10549-017-4199-3. Epub 2017 Mar 21. PMID 28324268